CLINICAL TRIAL: NCT02716233
Title: A French Protocol for the Treatment of Acute Lymphoblastic Leukemia (ALL) in Children and Adolescents
Acronym: CAALL-F01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P091205
Record Dates: First submitted 2016-02-15; First posted 2016-03-23 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): pegaspargase 2500 IU/m2 x 1: infusion of a conventional dose of pegaspargase during induction therapy: 2500 IU/m2x1
  Interventions: Drug: pegaspargase 2500 IU/m2 x 1
- Arm 2 (Experimental): pegaspargase 1250 IU/m2 x 2: fractionation of the 2500 IU/m2 pegaspargase dose in two infusions of 1250 IU/m2 each during delayed intensification
  Interventions: Drug: pegaspargase 1250 IU/m2 x 2

INTERVENTIONS:
Drug: pegaspargase 1250 IU/m2 x 2 — only for ALL of standard risk and medium risk
  Other Names: ONCASPAR 1250 IU/m2 x 2
  Arms: Arm 2
Drug: pegaspargase 2500 IU/m2 x 1 — only for ALL of standard risk and medium risk
  Other Names: ONCASPAR 2500 IU/m2 x 1
  Arms: Arm 1

SUMMARY:
A still major question in the field of acute lymphoblastic leukemia (ALL) in children - an extremely heterogeneous disease though curable in 80-90% of children and 70-80% of the adolescents - is the optimal use of L-asparaginase (ASNase). It is known that administering ASNase results in the depletion of asparagine circulating in the blood, which starves the leukemic cells and results in their death. But indeed the use of ASNase varies between protocols considering the different brands, the dose and the administration modalities. Oncaspar (PEGylated E. coli asparaginase, pegaspargase) was thus developed with the goal of reducing the immunogenicity of the native ASNase.

This is a French prospective multicentric cohort study of children and adolescents with ALL, stratified on (i) the type of ALL ( B vs T) and (ii) the anticipated risk (stratified in 3 groups for childhood B-cell precursor (BCP)-ALL and 2 groups for T-cell ALL).

It aims to answer to two different issues:

1. Randomized question: what is the best way to administer pegaspargase? A cohort of children and adolescents with standard or medium risk ALL will be randomized to receive during induction either one infusion of ONCASPAR® 2500 IU/m2 at D12 or two infusions of ONCASPAR® at 1250 IU/m2 each at D12 and D26. Patients will then receive 2500 IU/m2 or 1250 IU/m2 per dose during consolidation and delayed intensification according to the initial arm of randomization.
2. Non randomized question: In the High/Very High Risk groups, a non randomized intensification of the scheme of asparaginase administration is proposed during induction therapy: 2 infusions of 2500 IU/m2/day (D12 and D26) will be administered. All patients will receive 2500 IU/m2 per dose during consolidation and delayed intensifications.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents Age > 12 months but < 18 yearsB-lineage or T- lineage ALL
* Written informed consent obtained before day 8 of treatment

Non inclusion criteria:

* L3 (Burkitt's leukemia) (LMB type protocols)
* Mixed Phenotype Acute Leukemia (WHO criteria).
* Infant ALL (age ≤ 365 days (Interfant 06 protocol)
* Secondary leukemia
* Patients previously treated with chemotherapy (steroid exposed patients can be included and stratified according to Section 3.5) Known allergy to pegylated products
* Pregnancy. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant must have a negative serum pregnancy before inclusion and a reliable contraception except oral contraceptives. The contraception should be maintained throughout the study and for 3 months after treatment discontinuation.
* Known HIV positivity
* CNS thrombosis during Prophase

Exclusion Criteria:

* Ph+/BCR-ABL ALL (ESPhALL protocol)
* CNS thrombosis before D12

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2044 (Actual)
Dates: Start 2016-09-19; Primary Completion 2022-04 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adequate (> 100 IU/L) asparaginase activity measured in the plasma at day 33 of induction therapy | Day 33
  asparaginase activity > 100 IU/L
Incidence of directly asparaginase-related severe toxicities (Grade ≥ 3 as assessed by CTCAE v4.0) observed during induction therapy | Between Day 12 of induction and Day 8 of consolidation
  Incidence of severe toxicities (Grade ≥ 3) directly asparaginase-related (CNS thrombosis, pancreatitis, anaphylaxis, and hyperbilirubinemia) between Day 12 and Day 49 of treatment and anyway before Day 8 of consolidation

SECONDARY OUTCOMES:
Incidence of asparagine depletion measured in plasma by a concentration below the Limit of Quantification (LOQ) of 0.4 micromol/L | Day 33 of induction
Incidence of adequate (> 100 IU/L) asparaginase activity measured in the plasma at day 40 of induction therapy | Day 40 of induction
Incidence of asparagine depletion measured in plasma by a concentration below the Limit of Quantification (LOQ) of 0.4 micromol/L | Day 40 of induction
Incidence of antibodies against asparaginase, measured in serum | Day 4 of delayed intensification
Incidence of silent inactivation | First 6-9 months
  Silent inactivation or subclinical hypersensitivity is defined as a plasma PEGasparaginase activity level <100 IU/L at day 7+/- 1 or <20 IU/L at day 14 +/- 11 after administration in a patient without clinical symptoms of allergy
Percentage of patients without switch to Erwinia asparaginase | First 6-9 months
Percentage of patients receiving more than 95% of the intended dose of asparaginase | First 6-9 months
Morphological Complete Remission (CR) rates | Day 35-Day 42
  Assessed on the whole population or on subgroups (B-Lineage ALL, T-cell ALL).
Minimal Residual Disease (MRD) | Day 35-Day 42, Day 65-Day 105
  MRD will be assessed by Ig/T cell receptor (TCR)-based real-time quantitative (RQ)-polymerase chain reaction (PCR), assessed on the whole population or on subgroups (B-Lineage ALL, T-cell ALL).
  Assessed on the whole population or on subgroups (B-Lineage ALL, T-cell ALL).
Cumulative Incidence of relapses | 5 years
  Assessed on the whole population or on subgroups (B-Lineage ALL, T-cell ALL).
Cumulative Incidence of relapse according to site of relapse | 5 years
  Bone-Marrow (BM) relapses, central nervous system (CNS) relapses, gonadal relapses, combined relapses.
  Assessed on the whole population or on subgroups (B-Lineage ALL, T-cell ALL).
All other adverse events related to asparaginase | within the first 7 weeks (Day 49) of treatment and anyway before Day 8 of consolidation
  Drug-induced hyperglycemia or diabetes, coagulopathy, allergy Non CNS thrombosis Grade 1-2 Adverse Events (AE): pancreatitis, hyperbilirubinemia
Late adverse events related to asparaginase | after Day 49 of induction or anyway at Day 8 of consolidation or after

CONTACTS AND LOCATIONS:
Locations (28):
- France (28):
  - CHU, Amiens
  - CHU, Angers
  - CHRU, Besançon
  - CHU, Bordeaux
  - CHU, Brest
  - CHU, Caen
  - CHU, Clermont-Ferrand
  - CHU, Dijon
  - CHU, Grenoble
  - CHU, Lille
  - CHU, Limoges
  - Chu-Ihope, Lyon
  - CHU, Marseille
  - CHU, Montpellier
  - CHU, Nancy
  - CHU, Nantes
  - CHU, Nice
  - CHU Saint Louis, Paris
  - CHU Armand Trousseau, Paris
  - CHU Robert Debré, Paris
  - CHU, Poitiers
  - CHU, Reims
  - CHU, Rennes
  - CHU, Rouen
  - CHU, Saint-Etienne
  - CHU, Strasbourg
  - CHU, Toulouse
  - CHU, Tours

IPD SHARING:
Plan to Share IPD: Undecided